CLINICAL TRIAL: NCT02463123
Title: Resting Energy Expenditure in Cardiac Patients Operated Under Cardiopulmonary Bypass
Brief Title: Energy Expenditure Estimation in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Efremov Sergey, anestesiologist, Meshalkin Research Institute of Pathology of Circulation
Other Study IDs: 01.2015
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Surgical Procedures; Intensive Care
MeSH Terms: interventions — Calorimetry, Indirect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Indirect calorimetry — Resting energy expenditure will be studied using indirect calorimeter CCM Express (Medgraphics Inc, USA).

SUMMARY:
Estimation of energy requirements is essential for adequate nutritional support in ICU. Indirect calorimetry being the golden standard of resting energy expenditure estimation is not available in most intensive care units. Different predictive equations have been developed, but not evaluated in cardiac population and have low accuracy in compare to the indirect calorimetry. The aim of present study is to develop cardio-specific equation for resting energy expenditure estimation.

ELIGIBILITY:
Inclusion Criteria:

* Patient of cardiothoracic ICU

Exclusion Criteria:

* Shock
* patients on ECMO
* Hypoxemia <60 mmHg
* Active bleeding
* Ventilation with FiO2 >0.6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after cardiothoracic interventions using cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure measured in kcal/day using indirect calorimetry | participants will be followed for the duration intensive care unit stay, an expected average 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Background] Efremov SM, Talaban VO, Ponomarev DN, Vedernikov PE, Chechenin MG, Artemieva VV, Lomivorotov VV. Development and Validation of a New Cardio-Specific Resting Energy Expenditure Equation for Adults. JPEN J Parenter Enteral Nutr. 2018 May;42(4):702-708. doi: 10.1177/0148607117711648. Epub 2017 Dec 19. PMID 28575581